CLINICAL TRIAL: NCT02805543
Title: The Correlation Between the Retrobulbar Hemodynamics and Intrarenal Hemodynamics in T2DM Patients During the Early Period
Status: Completed | Type: Observational
Sponsor: Fourth People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Jin-song Kuang, Chief physician, Fourth People's Hospital of Shenyang
Other Study IDs: 20160204; F11-262-9-25 (Other Grant/Funding Number: Natural Science Foundation of Shenyang)
Record Dates: First submitted 2016-06-12; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- diabetes group: 34 T2DM patients without vascular complications as diabetes group
  Interventions: Device: Color doppler imaging
- control group: 32 healthy people were recruited as control group
  Interventions: Device: Color doppler imaging

INTERVENTIONS:
Device: Color doppler imaging

SUMMARY:
Objective: The main target of this study was to research the early changes of retrobulbar and intrarenal hemodynamics, then to research the correlation between them in type 2 diabetes (T2DM) patients without diabetic kidney disease (DKD) and diabetic retinopathy (DR).

Method: 35 T2DM patients (diabetes group) without vascular complications and 30 healthy people (control group) were recruited to research the early changes of renal function, retrobulbar and intrarenal hemodynamics, and then to research the correlation between them. The primary endpoints were the intrarenal hemodynamic (bilateral kidney RI) in bilateral interlobular renal arteries were evaluated using Doppler Sonographic; the secondary endpoints were the retrobulbar hemodynamics RI in the bilateral central retinal artery (CRA), posterior ciliary artery (PCA), and arteria ophthalmica (OA) were evaluated using color doppler imaging (CDI); the tertiary endpoints were the biochemical endpoints: blood-fat (TC, HDL-C, LDL-C, and TG), FPG, 2hPG, HbA1c, and renal function parameters (BUN, Cr, and GFR); in addition, the albumin excrete rate (AER), urinary albumin/creatinine ratio (UACR) were measured.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were diagnosed with T2DM according to the guidelines of the American Diabetes Association ;
2. No smoking history, pulmonary disease, cold, nor pulmonary infection within a fortnight;
3. Did not have hepatopathy, nephropathy, hyperuricemia, and gastrointestinal disease; and
4. Likely to have good compliance and able to visit our hospital for periodic assessments.

Exclusion Criteria:

1. T1DM, gestation and lactation;
2. Renal inadequacy,hypohepatia,and heart failure;
3. Intensive care with insulin treatment;
4. The patients combined with DR and hypertension (antihypertensive drugs were used);
5. Patients with other eye conditions that could affect the blood flow, such as high degree myopia, maculopathy of any origin, glaucoma, and those with a history of laser treatment or intraocular surgery;
6. The patients combinated with DKD;
7. Patients with other renal conditions that could affect the blood flow, such as urolithiasis, urinary infection, and renal cyst (diameter > 3 cm);
8. Cholesterol-lowering drugs can not control the blood-fat (TC > 250 mg/dl, HDL-C < 30 mg/dL, LDL-C > 170 mg/dl, TG > 200 mg/dl) adequately.

Ages: 35 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators selected 45 T2DM patients (25 males, 20 females) without microangiopathy (DR and DKD) as diabetes group and 38 healthy people (21 males, 17 females) as control group from the diabetic outpatient clinic in Shenyang the Fourth Hospital of People, but only 34 patients (19 males, 15 females) in the diabetes group and 32 healthy people (17 males, 15 females) can be researched in our study, all the participants were the Chinese Hans. All patients were provided a diet and exercise program by professional nutritionists.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Intrarenal hemodynamic (bilateral kidney RI) in bilateral interlobular renal arteries were evaluated using Doppler Sonographic in 34 patients | 3 weeks
  RI(resistivity index)
Retrobulbar RI in the bilateral Retrobulbar artery were evaluated using color doppler imaging (CDI) in 34 patients | 3 weeks
  RI(resistivity index),Retrobulbar artery［central retinal artery (CRA), posterior ciliary artery (PCA), and arteria ophthalmica (OA)］
The correlation between the bilateral retrobulbar RI and bilateral kidney RI in 34 patients | 3 weeks
  RI(resistivity index)